CLINICAL TRIAL: NCT06946550
Title: 1470 nm Non-Ablative Laser for the Treatment of Scarring Alopecia: A Clinical and Mechanistic Study
Brief Title: Non-Ablative Laser to Treat Scarring Alopecia With Hair Follicle Gene Expression Analysis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Sciton (Industry); American Society for Laser Surgery and Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-16805
Record Dates: First submitted 2025-04-19; First posted 2025-04-27 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Scarring Alopecia
Keywords: alopecia; laser
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Scarring alopecia (Experimental): Patients with scarring alopecia will receive 3 treatments with the non-ablative Sciton HALO laser (1470nm). Each laser treatment will take approximately 10 to 15 minutes per subject.
  Interventions: Device: 1470nm non-ablative fractional laser

INTERVENTIONS:
Device: 1470nm non-ablative fractional laser — Patients with scarring alopecia will be treated with the non-ablative Sciton HALO laser (1470nm).

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of a non-ablative 1470 nm laser in treating scarring alopecia in adults. The study will also investigate the biochemical molecular pathways involved in laser therapy by analyzing hair follicle gene expression before and after laser treatment.

The main questions it aims to answer are:

1. Does a non-ablative laser work to effectively treat scarring alopecia?
2. What molecular pathways are associated with the laser's effects on hair follicles in scarring alopecia?

Participants with scarring alopecia will:

* Receive 3 laser treatments, spaced 1 month apart (Month 1, Month 2, Month 3), and attend 5 follow-up visits (Month 4, Month 6, Month 9, Month 12 and Month 15)
* Have hair follicle samples collected via hair plucking of 10 hairs prior to the start and 1-month post-completion of laser treatments for gene expression analysis of inflammatory and fibrosis pathways implicated in scarring alopecia. Hair samples will be de-identified and kept anonymous.
* Fill out questionnaires at each visit
* Keep a diary of any side effects from laser treatments

DETAILED DESCRIPTION:
This is a prospective, single-center, open-label, baseline-controlled study evaluating the molecular pathways of the effects of a non-ablative 1470 nm laser for the treatment of scarring alopecia. 5 treatment-naive (or at least 1 year since last hair loss medical treatment) participants with prior biopsy-proven or clinically diagnosed scarring alopecia will be enrolled into the study. Hair follicle samples will be obtained via hair plucking prior to the first laser treatment (Month 1) and 1-month post-completion of the laser treatments (Month 4). Each subject will receive 3 laser treatments, spaced 1 month apart, and 5 follow-up visits, planned for Month 4, Month 6, Month 9, Month 12 and Month 15. Measurement outcomes will be compared to baseline.

For this study, the investigators will use the non-ablative Sciton HALO ® laser (1470nm). The non-ablative fractionated treatments with minimal downtime provide synergistic benefit of minimizing tissue damage while improving treatment tolerance and efficiency. The laser works by creating micro-channels in the dermis of the pilosebaceous unit, while leaving bridges of untouched tissue for improved permeability, faster healing, and enhanced delivery of topical treatments. The laser creates controlled zones of coagulation within the dermis. The parameters of the laser will be set according to optimal operation protocol and in accordance with guidelines set forth by Sciton and standard of care. Each laser treatment will take approximately 10 to 15 minutes per subject. Pre-treatment procedure will consist of the application of topical anesthetic then cleaning of the affected area of the scalp with antiseptic, either 70% ethanol or 3% hydrogen peroxide. Post-treatment care will follow standard of care. The U.S. Food and Drug Administration (FDA) has cleared the 1470 nm laser for dermatologic purposes. This study will use the laser off-label for the treatment of alopecia. This laser has been approved for the treatment of skin resurfacing; however, research on the use of this laser in alopecia is lacking.

The investigator team plans to define the molecular mechanisms involved in laser treatment of scarring alopecia. Using a non-invasive method of hair plucking, we will evaluate the hair follicle gene expression of inflammatory and fibrosis pathways in participants with scarring alopecia prior to treatment. Changes in gene expression through gene expression analysis of hair follicles at 1-month post-laser treatment completion will also be identified.

The follow up phase will consist of clinical assessments including before and after photographs graded by blinded observers and hair density evaluation using the Canfield HairMetrix ® device. Subjects are instructed to inform clinical staff after the treatment if any adverse events are experienced and will complete patient questionnaires, pain scores, and self-assessments of hair growth.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, at least 18 years of age at time of informed consent, seeking treatment for scarring alopecia
* Subject must be able to read, understand, and voluntarily sign and date an IRB-approved informed consent form
* Subjects with biopsy-proven or clinically diagnosed scarring alopecia recorded within the past 6 months. An established clinical diagnosis will be confirmed by a licensed dermatologist as in previously published hair plucking studies (eg. using trichoscopy and a positive pull test). Subjects must have a stable hair loss treatment regimen with a plateau in results for at least 3 months.
* Subject agrees to not make any changes to their daily hair treatment regimen or start any medications for hair loss such as minoxidil during the study.
* Subjects able and willing to comply with the treatment protocol and follow-up schedule and requirements.
* Understands and accepts the obligation not to undergo any other procedures in the areas to be treated throughout the follow-up period.

Exclusion Criteria:

* Subject does not have capacity to consent to the study
* No ethnic or racial group restrictions
* Subject does not have scarring alopecia
* History of intralesional steroid injections to the scalp in the last 12 months
* Pregnant Women
* Any medical condition that in the consideration of the investigator, would present an increased risk of a photosensitivity reaction to the subject.
* Any previous hospitalization or surgical procedure in the treatment area in the past 12 months, or major surgery in the last 6 months.
* Allergy or history of prior reaction to lidocaine
* History of immunosuppression/immune deficiency disorders (including AIDS and HIV infection), and/or any history of systemic chemotherapy in the prior 12 months.
* Recent COVID-19 infection
* History or current use of the following prescription medications:
* Immunosuppressive medications/biologics, 6 months prior to and during the study
* Accutane or other systemic retinoids within the past twelve months
* Smoking or vaping in the past 12 months.
* History of uncontrolled hyperlipidemia, uncontrolled diabetes mellitus, uncontrolled hepatitis, or uncontrolled bleeding disorders.
* History of major depressive disorders or uncontrolled endocrine disorders including but not limited to; hypothyroidism, Hashimoto's thyroiditis, or hyperthyroidism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Clinician Global Aesthetic Improvement Scale | Month 2, Month 3, Month 4, Month 6, Month 9, Month 12, Month 15
  A clinician will answer the following question after evaluating baseline photos and current photos (at each specified point in time).
  Please choose the option that better represents the change in hair growth in the treatment area.
  The options will be as follows: -3 = Greatly worsened -2 = Moderately worsened -1 = Slightly worsened 0 = No change 1 = Slightly worsened 2 = Moderately improved 3 = Greatly improved. Higher scores will be associated with improved hair growth in treatment area as assessed by a clinician. Group scores will be summarized by each specified point in time.
Subject Global Aesthetic Improvement Scale | Month 2, Month 3, Month 4, Month 6, Month 9, Month 12, Month 15
  Subjects will answer the following questions after evaluating baseline photos and current photos (at each specified point in time).
  Please choose the option that better represents the change in hair growth in each treatment area from baseline to today.
  The options will be as follows: -3 = Greatly worsened -2 = Moderately worsened -1 = Slightly worsened 0 = No change 1 = Slightly improved 2 = Moderately improved 3 = Greatly improved, such that higher scores are associated with the subjects' self-assessment of improved aesthetic for each assessment. Group scores will be summarized by each specified point in time.
Hair density | Baseline/Month 1, 2, 3, 4, 6, 9, 12, 15
  Hair density assessed using Canfield HairMetrix imaging device measured as average number of hairs (as reported by the device) per follicular unit for each treatment area (patient-dependent).
Hair counts | Baseline/Month 1, 2, 3, 4, 6, 9, 12, 15
  Hair counts assessed using Canfield HairMetrix imaging device measured as average hair count per square centimeter (as reported by the device) per treatment area (patient-dependent).

SECONDARY OUTCOMES:
Subject Satisfaction Questionnaire | Month 2, Month 3, Month 4, Month 6, Month 9, Month 12, Month 15
  Comparing baseline photos and current photos of the scalp, the participant will answer the following questions:
  1. Please choose the option that best represents the change in how your hair looks OVERALL in the area treated? 2. Please choose the option that best represents the change in your hair THICKNESS in the area treated? 3. Please choose the option that best represents the change in your hair SHEDDING/LOSS in the area treated? 4. Please choose the option that best represents the change in your hair DARKNESS in the area treated.
  The options will be: -3 = Greatly worsened -2 = Moderately worsened -1 = Slightly worsened 0 = No change 1 = Slightly improved 2 = Moderately improved 3 = Greatly improved.
  The average values will be reported for each specified point in time for each of the 4 parameters (overall, thickness, shedding/loss, and darkness). Only the first 4 questions of the subject satisfaction questionnaire (as specified above) are considered relevant to the outcome.
Change in Dermatology Life Quality Index | From Baseline/Month 1 to Month 15
  The participant will answer a series of 10 questions to measure how much their scarring alopecia has affected their life over the past week. It uses a 10-question self-administered questionnaire where each question is scored from 0 to 3, with a total score ranging from 0 to 30. The change from baseline/Month 1 to the end of the study (Month 15) will be summarized. Positive scores will be indicative of greater impact on the quality of life and negative scores will be indicative of reduced impact on the quality of life.

OTHER OUTCOMES:
Hair follicle inflammatory and fibrosis pathway gene expression analysis | Hair plucking to obtain hair follicle samples will be performed Month 1 (prior to the start of laser treatments) and Month 4 (1-month post completion of laser treatments)
  Subjects will undergo hair plucking twice-once prior to treatment and once more at the 1-month follow-up of the study. Ten hairs will be plucked from scalp and placed immediately into a buffer solution in a de-identified tube. The procedure will take three minutes and will have no lasting side effects. Ribonucleic acid (RNA) will then be extracted, reverse-transcribed to complementary DNA (cDNA), and sequenced. Bioinformatic analysis will be done using Kallisto and DESeq2 software median-of-ratios method. A single unit of measurement (eg., log₂ fold-change or normalized counts) will be used to report all genes of interest, mainly inflammatory and fibrosis pathways implicated in scarring alopecia (eg. -TGF-β1, NLRP3, IL-1β, IL-18, COL1A1, COL3A1, CTGF, CCL2, CCL21, CXCL6).

CONTACTS AND LOCATIONS:
Overall Officials: Kseniya Kobets, MD, Principal Investigator — Albert Einstein College of Medicine Montefiore Medical Center
Locations (1):
- Montefiore Einstein Advanced Care, Elmsford, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Karnik P, Tekeste Z, McCormick TS, Gilliam AC, Price VH, Cooper KD, Mirmirani P. Hair follicle stem cell-specific PPARgamma deletion causes scarring alopecia. J Invest Dermatol. 2009 May;129(5):1243-57. doi: 10.1038/jid.2008.369. Epub 2008 Dec 4. PMID 19052558
- [Background] Anzai A, Wang EHC, Lee EY, Aoki V, Christiano AM. Pathomechanisms of immune-mediated alopecia. Int Immunol. 2019 Jul 13;31(7):439-447. doi: 10.1093/intimm/dxz039. PMID 31050755
- [Background] Hordinsky M. Scarring Alopecia: Diagnosis and New Treatment Options. Dermatol Clin. 2021 Jul;39(3):383-388. doi: 10.1016/j.det.2021.05.001. PMID 34053592
- [Background] Van Mater D, Kolligs FT, Dlugosz AA, Fearon ER. Transient activation of beta -catenin signaling in cutaneous keratinocytes is sufficient to trigger the active growth phase of the hair cycle in mice. Genes Dev. 2003 May 15;17(10):1219-24. doi: 10.1101/gad.1076103. PMID 12756226
- [Background] Jamerson TA, Conover Talbot C Jr, Dina Y, Kwatra SG, Garza LA, Aguh C. Gene expression profiling suggests severe, extensive central centrifugal cicatricial alopecia may be both clinically and biologically distinct from limited disease subtypes. Exp Dermatol. 2022 May;31(5):789-793. doi: 10.1111/exd.14524. Epub 2022 Jan 20. PMID 35007355
- [Background] Tanakol A, Oba MC, Uzuncakmak TK, Askin O, Kutlubay Z. Treatment of alopecia areata with 2940-nm fractional erbium:yttrium-aluminum-garnet laser. Dermatol Ther. 2020 Nov;33(6):e13978. doi: 10.1111/dth.13978. Epub 2020 Aug 6. PMID 32633447
- [Background] Cho SB, Goo BL, Zheng Z, Yoo KH, Kang JS, Kim H. Therapeutic efficacy and safety of a 1927-nm fractionated thulium laser on pattern hair loss: an evaluator-blinded, split-scalp study. Lasers Med Sci. 2018 May;33(4):851-859. doi: 10.1007/s10103-018-2437-5. Epub 2018 Jan 16. PMID 29340854
- [Background] Ke J, Guan H, Li S, Xu L, Zhang L, Yan Y. Erbium: YAG laser (2,940 nm) treatment stimulates hair growth through upregulating Wnt 10b and beta-catenin expression in C57BL/6 mice. Int J Clin Exp Med. 2015 Nov 15;8(11):20883-9. eCollection 2015. PMID 26885014
- [Background] Raffi J, Suresh R, Agbai O. Clinical recognition and management of alopecia in women of color. Int J Womens Dermatol. 2019 Aug 22;5(5):314-319. doi: 10.1016/j.ijwd.2019.08.005. eCollection 2019 Dec. PMID 31909150
- [Background] Jimenez F, Izeta A, Poblet E. Morphometric analysis of the human scalp hair follicle: practical implications for the hair transplant surgeon and hair regeneration studies. Dermatol Surg. 2011 Jan;37(1):58-64. doi: 10.1111/j.1524-4725.2010.01809.x. Epub 2010 Nov 11. PMID 21070465
- [Background] Savoia A, Accardo C, Vannini F, Di Pasquale B, Baldi A. Outcomes in thread lift for facial rejuvenation: a study performed with happy lift revitalizing. Dermatol Ther (Heidelb). 2014 Jun;4(1):103-14. doi: 10.1007/s13555-014-0041-6. Epub 2014 Jan 17. PMID 24436079
- [Background] Shimojima K, Hashimoto M, Yamaoka Y, Kapoor KM. Combination Treatment with Cryolipolysis and Hyaluronic Acid Fillers for Jawline Enhancement. Clin Cosmet Investig Dermatol. 2024 Dec 20;17:2989-2998. doi: 10.2147/CCID.S492091. eCollection 2024. PMID 39723342
- [Background] Tsur Shenhav L, Shehade W, Muravnik G, Horovitz T, Artzi O. The Safety and Efficacy of a Dual CO 2 and 1570-nm Hybrid Laser for Periorbital Rejuvenation. Dermatol Surg. 2023 May 1;49(5):479-482. doi: 10.1097/DSS.0000000000003750. Epub 2023 Mar 6. PMID 36877122
- [Background] Constantinou A, Polak-Witka K, Tomazou M, Oulas A, Kanti V, Schwarzer R, Helmuth J, Edelmann A, Blume-Peytavi U, Spyrou GM, Vogt A. Dysbiosis and Enhanced Beta-Defensin Production in Hair Follicles of Patients with Lichen Planopilaris and Frontal Fibrosing Alopecia. Biomedicines. 2021 Mar 7;9(3):266. doi: 10.3390/biomedicines9030266. PMID 33800045
- [Background] Sanchez P, Serrano Falcon C, Martinez Rodriguez S, Torres JM, Serrano S, Ortega E. mRNA Levels of Aromatase, 5alpha-Reductase Isozymes, and Prostate Cancer-Related Genes in Plucked Hair from Young Men with Androgenic Alopecia. Int J Mol Sci. 2023 Dec 14;24(24):17461. doi: 10.3390/ijms242417461. PMID 38139289
- [Background] Bray NL, Pimentel H, Melsted P, Pachter L. Near-optimal probabilistic RNA-seq quantification. Nat Biotechnol. 2016 May;34(5):525-7. doi: 10.1038/nbt.3519. Epub 2016 Apr 4. PMID 27043002
- [Background] Aguh C, Dina Y, Talbot CC Jr, Garza L. Fibroproliferative genes are preferentially expressed in central centrifugal cicatricial alopecia. J Am Acad Dermatol. 2018 Nov;79(5):904-912.e1. doi: 10.1016/j.jaad.2018.05.1257. Epub 2018 Jun 18. PMID 29913259